CLINICAL TRIAL: NCT01283126
Title: Blood/Interstitial Glucose Measurements and Cognitive Function During Hypoglycemia and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHS #: 2010-09
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia, cognitive function
MeSH Terms: conditions — Hypoglycemia | interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Euglycemic and hypoglycemic clamp (Experimental): Subjects will complete clamp study visit.
  Interventions: Procedure: euglycemic and hypoglycemic clamp

INTERVENTIONS:
Procedure: euglycemic and hypoglycemic clamp — Subjects will undergo standard euglycemic and hypoglycemic clamps, and will have concurrent assessments of cognitive function and measurement of interstitial glucose concentrations.
  Other Names: clamp

SUMMARY:
The purpose of this study is to find out the effects of hypoglycemia on cognition in healthy individuals and how well changes in (interstitial) tissue glucose levels correlate with changes in cognitive function as compared to blood glucose levels.

DETAILED DESCRIPTION:
Subjects will undergo hypoglycemic clamps during which interstitial glucose will be measured and cognitive function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* non obese (BMI <30), ages 18-50

Exclusion Criteria:

* renal or hepatic failure
* cancer or lymphoma
* malabsorption or malnourishment
* hypercortisolism
* alcoholism or drug abuse
* anemia
* eating disorder or depression
* coronary artery disease
* Arrhythmias
* hypertension
* on medications known to affect the blood glucose to be measured such as
* glucocorticoids
* on blood thinning agents

  * Pregnant women, breastfeeding women and women who want to become pregnant in the next 6 months will be excluded from the study.
  * Subjects who have donated blood two weeks prior to the study.
  * Allergies to pig derived products (Heparin will be used)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
cognitive function correlation to blood or interstitial glucose | 1 year
  This investigator initiated study will evaluate cognitive function at the onset, during and following recovery from hypoglycemia and will determine if cognitive function correlates better with blood or interstitial glucose concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Joslin Diabetes Center; Greeshma K Shetty, MD, Study Chair — Joslin Diabetes Center; Gail Musen, PhD, Study Chair — Joslin Diabetes Center; Gail Adler, MD, PhD, Study Chair — Brigham and Women's Hospital
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No